CLINICAL TRIAL: NCT00137384
Title: The Role of Cortical Coherence in Focal Hand Dystonia
Brief Title: Movement-Related Brain Networks Involved in Hand Dystonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050228; 05-N-0228
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04-27

CONDITIONS: Movement Disorder; Focal Dystonia
Keywords: Magnetoencephalogram; Functional Connectivity; Electroencephalogram (EEG); Focal Hand Dystonia; Spectral Analysis; Healthy Volunteer; HV
MeSH Terms: conditions — Movement Disorders; Dystonic Disorders; Dystonia, Focal, Task-Specific

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will use various methods to measure the activity of the motor cortex (the part of the brain that controls movements) in order to learn more about focal hand dystonia. Patients with dystonia have muscle spasms that cause uncontrolled twisting and repetitive movement or abnormal postures. In focal dystonia, just one part of the body, such as the hand, neck or face, is involved.

Patients with focal hand dystonia and healthy normal volunteers between 18 and 65 years of age may be eligible for this study. Each candidate is screened with a medical history, physical examination and questionnaire. Participants undergo the following procedures:

Finger Movement Tasks

Subjects perform two finger movement tasks. In the first part of the study, they move their index finger repetitively from side to side at 10-second intervals for a total of 200 movements in four blocks of 50 at a time. In the second part of the study, subjects touch their thumb to the other four fingers in sequence from 1, 2, 3 and 4, while a metronome beats 2 times per second to help time the movements. This sequence is repeated for a total of 200 movements in four blocks of 50 at a time.

Electroencephalography

This test records brain waves. Electrodes (metal discs) are placed on the scalp with an electrode cap, a paste or a glue-like substance. The spaces between the electrodes and the scalp are filled with a gel that conducts electrical activity. Brain waves are recorded while the subject performs a finger movement task, as described above.

Magnetoencephalography

MEG records magnetic field changes produced by brain activity. During the test, the subjects are seated in the MEG recording room and a cone containing magnetic field detectors is lowered onto their head. The recording may be made while the subject performs a finger task.

Electromyography

Electromyography (EMG) measures the electrical activity of muscles. This study uses surface EMG, in which small metal disks filled with a conductive gel are taped to the skin on the finger.

Magnetic resonance imaging

MRI uses a magnetic field and radio waves to produce images of body tissues and organs. The patient lies on a table that can slide in and out of the scanner (a narrow metal cylinder), wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning. Most scans last between 45 and 90 minutes. Subjects may be asked to lie still for up to 30 minutes at a time, and can communicate with the MRI staff at all times during the procedure.

Questionnaire

This questionnaire is designed to detect any sources of discomfort the subject may have experienced during the study.

DETAILED DESCRIPTION:
Objective

Dystonia is a disabling movement disorder that manifests with sustained co-contraction of agonist and antagonist muscles, giving rise to abnormal twisted postures and overflow of muscle activity. Abnormal neurophysiologic parameters of the somatosensory and motor cortex have been demonstrated, although it is unclear how these changes lead to the predominant motor manifestations. In normal voluntary movement, communication between sensory and motor cortices is important and these interactions may be dysfunctional in dystonia. Coherence is a powerful method used to assess brain communication and has been instrumental in demonstrating the interregional interactions involved in normal movement. Inappropriate connectivity in terms of the duration of communication or the extent of spread over sensorimotor areas may give rise to the involuntary overflow of movements that characterize dystonia. We propose to examine changes in coherence associated with disorganized movements to yield insight as to the brain networks involved in the development and expression of the disease.

Study population

Patients with focal hand dystonia and normal volunteers will take part in the study.

Design

In this study, EEG/MEG coherence analysis will be used to investigate corticocortical and corticomuscular interactions during voluntary hand movements in focal hand dystonia patients and normal subjects. Power spectral changes in the beta and alpha frequency range over the hand sensorimotor cortex will be studied using a 28-channel EEG montage while subjects perform various tasks involving the hand. The interregional coherence between sensory and motor, premotor and motor, and interhemispheric cortices will be assessed for changes between study populations.

Outcome Measures

Comparison of interregional coherence changes will be performed between dystonia patients and normal volunteers as well as between affected and unaffected sides. Furthermore, coherence changes will be compared between rest and during task performance.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Normal subjects: Healthy volunteers ages 18 and older who consent to participate in the study
* Patients ages 18 and older diagnosed with focal hand dystonia unilateral focal hand dystonia who consent to participate in the study

EXCLUSION CRITERIA:

* Normal subjects: abnormal neurologic exam or history of previous neurological disease that might affect the functioning of the hands
* Dystonia patients: presence of a second neurologic disease or condition that might affect the functioning of the hands; abnormal neurologic findings on exam not related to the focal hand dystonia that might affect the functioning of the hands; the use of Botulinum toxin within 3 months prior to study participation
* For MRI studies, patients with metallic implants will be excluded to avoid potential risks from this procedure
* For MRI studies, women who are pregnant are excluded from this part of the protocol. All women of childbearing potential will have a pregnancy test performed prior to MRI studies, which must be negative, before proceeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-08-25; Study Completion 2018-04-27

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abbruzzese G, Berardelli A. Sensorimotor integration in movement disorders. Mov Disord. 2003 Mar;18(3):231-240. doi: 10.1002/mds.10327. PMID 12621626
- [Background] Abbruzzese G, Marchese R, Buccolieri A, Gasparetto B, Trompetto C. Abnormalities of sensorimotor integration in focal dystonia: a transcranial magnetic stimulation study. Brain. 2001 Mar;124(Pt 3):537-45. doi: 10.1093/brain/124.3.537. PMID 11222454
- [Background] Andres FG, Gerloff C. Coherence of sequential movements and motor learning. J Clin Neurophysiol. 1999 Nov;16(6):520-7. doi: 10.1097/00004691-199911000-00004. PMID 10600020